CLINICAL TRIAL: NCT00072813
Title: MRI in Autosomal Dominant Partial Epilepsy With Auditory Features
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040033; 04-N-0033
Record Dates: First submitted 2003-11-10; First posted 2003-11-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-11-12

CONDITIONS: Epilepsies, Partial
Keywords: Genetics; Seizures; Brain Imaging; Diffusion; Temporal Lobe
MeSH Terms: conditions — Epilepsies, Partial; Seizures

SUMMARY:
This study will examine the possible structural and functional abnormalities in patients with an inherited form of epilepsy. It will use magnetic resonance imaging (MRI). Uncontrolled epilepsy is a serious neurological problem with major harmful medical, social, and psychological effects, as well as greater mortality compared with the general population. The cost per year in the United States is at least $12.5 billion. There have been advances in diagnosing the disease, but the cause cannot be determined in many cases. Recently, several seizure syndromes found in families have been described. One syndrome of particular interest involves the lateral temporal lobe of the brain and often includes auditory features. Patients with that kind of syndrome may hear monotonous unformed sounds, but sometimes they may hear complex sounds, such as a song.

Patients are eligible for this study if they have a specific form of familial epilepsy that is being studied at Columbia University in New York. Family members without seizures are eligible as well. All the patients in the study will be evaluated at Columbia before participating. Healthy volunteers aged 18 to 55 also may be eligible for this study.

Participants will undergo a medical history and physical examination. During the study, they may have three or four sessions of MRI. During the MRI, patients will lie still on a table that can slide in and out of a metal cylinder surrounded by a strong magnetic field. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. Patients may be asked to lie still for up to 60 minutes at a time. As the scanner takes pictures, there will be loud knocking noises, and the patients will wear earplugs to muffle the sound. Patients will be able to communicate with the MRI staff at all times during the scan and may ask to be moved out of the machine at any time. Some scans may be done in a 3 Tesla scanner. It is the latest advance in MRI, with a stronger magnetic field than in the more common 1.5 Tesla scanner. Functional MRI (fMRI) is done while patients are performing tasks, such as moving a limb or speaking. Patients will have an opportunity to practice such tasks before entering the scanner. The fMRI will take about 1 hour.

...

DETAILED DESCRIPTION:
Objectives: to study potential structural and functional abnormalities in patients with an inherited form of epilepsy.

Study Population: Patients with autosomal dominant partial epilepsy with auditory features, a newly described syndrome, asymptomatic family members who are gene carriers, and unaffected family members, and normal volunteers.

Design: magnetic resonance imaging, electroencephalography, and magnetoencephalography.

Outcome measures: detection of structural lesions; regional activation patterns on fMRI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients and family members in kindreds with ADPEAF evaluated by Dr. Ruth Ottman at CPMC:

14 patients with seizures and the LGl1 mutation.

14 family members with the mutation but no seizures.

14 Non-affected family members, who are not carriers of the LGl1 mutation.

30 normal controls selected at NIH, and screened in the CES outpatient clinic with a physical and neurological examination.

EXCLUSION CRITERIA:

Subjects unable or unwilling to undergo MRI, EEG, and MEG.

Women who are pregnant.

Subjects under 18.

Subjects with medical conditions other than ADPEAF that may affect brain function.

Subjects taking medications or neuroactive substances that may affect brain function.

Healthy volunteers must be below the age of 55, to reduce the chance of vascular chnages that could affect MRI.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2003-11-10; Primary Completion 2009-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Columbia University, New York, New York

REFERENCES:
- [Background] Baker GA, Nashef L, van Hout BA. Current issues in the management of epilepsy: the impact of frequent seizures on cost of illness, quality of life, and mortality. Epilepsia. 1997;38 Suppl 1:S1-8. doi: 10.1111/j.1528-1157.1997.tb04511.x. PMID 9092951
- [Background] Bastos AC, Korah IP, Cendes F, Melanson D, Tampieri D, Peters T, Dubeau F, Andermann F. Curvilinear reconstruction of 3D magnetic resonance imaging in patients with partial epilepsy: a pilot study. Magn Reson Imaging. 1995;13(8):1107-12. doi: 10.1016/0730-725x(95)02019-p. PMID 8750323
- [Background] Bastos AC, Comeau RM, Andermann F, Melanson D, Cendes F, Dubeau F, Fontaine S, Tampieri D, Olivier A. Diagnosis of subtle focal dysplastic lesions: curvilinear reformatting from three-dimensional magnetic resonance imaging. Ann Neurol. 1999 Jul;46(1):88-94. doi: 10.1002/1531-8249(199907)46:13.0.co;2-4. PMID 10401784